CLINICAL TRIAL: NCT05746364
Title: Case-Series Examination of a Brief CAT-Informed Intervention for Young People Experiencing Difficulties With Eating (RIDE)
Acronym: RIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Peter Taylor, Senior clinical lecturer, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS002023
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIDE intervention (Experimental): Cognitive analytic therapy (CAT)-informed brief therapy for young people struggling with disordered eating
  Interventions: Behavioral: Brief CAT-Informed Intervention for Young People experiencing Difficulties with Eating

INTERVENTIONS:
Behavioral: Brief CAT-Informed Intervention for Young People experiencing Difficulties with Eating — The therapy draws upon the principles of Cognitive Analytic Therapy (CAT), focussing on collaboratively identifying relational patterns (relationships with self and others) that young people experience difficulties with. The young person will be invited to attend 5 weekly sessions, each lasting 30-50 minutes. It will be delivered within a seven-week window (allowing for cancellations/missed sessions). Researchers will follow the RIDE manual treatment guide, which was developed by Clinical Psychologists, CAT accredited therapists and researchers.

SUMMARY:
Eating Disorders (ED) are mental health conditions where people alter food intake in some way to help with weight gain, managing emotions or other situations. EDs are increasingly common in young people. They can cause both the young person and those around them significant distress. Talking therapies can help.

Cognitive Analytic Therapy (CAT) is a talking therapy that is becoming increasingly widely used within the NHS to help with a wide range of problems. CAT focuses on the relationships clients have with themselves and others around them. From CAT, we have developed Relational Intervention for Difficulties with Eating (RIDE), This is a brief talking therapy. The aim is to help the young person and those around them build an understanding of their difficulties. This will hopefully mean others can support them with their disordered eating.

The aim of the study is to examine the feasibility (is it possible to conduct a study about this intervention?) and acceptability (do participants find the therapy is helpful and makes sense to them?) of RIDE. As a secondary aim, the study will look at whether RIDE shows preliminary evidence for positive change on relevant measures of psychological difficulties (e.g. distress, how young people feel about themselves and others).

The study will aim to recruit nine young people (aged between 14-25) with ED. Participants must be under the care of an ED service. They will attend 8 appointments (3 assessment, 5 therapy) either at their home, University of Manchester campus or a health service clinic. A video conferencing platform (e.g. Zoom, Teams) can be used if required. Participants will complete questionnaires before, during and after therapy.

The findings will help to develop the therapy and improve further testing in larger studies. If successful, RIDE could be available as a treatment for young people.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be between the ages of 14 - 25 years.
* Participants will be under the care of a mental health team and have a clinician allocated to them within local ED Services.

Exclusion Criteria:

* Young people will be excluded if they are currently receiving alternative one-to-one psychological therapy (not including family interventions or skill-based groups).
* Young people will be excluded if they have a moderate to severe intellectual disability which would impair their ability to participate without considerable adaptations being made to the intervention, as judged by the young person or the clinical team.
* Young people will be excluded if they have inadequate English-language speaking skills due to limitations in their ability to engage with talking therapies in the English language.
* Young people will be excluded if they are judged at high risk of harm to themselves, operationalised as having current suicidal thoughts with a high intent or active plan to end their life. This includes individuals who are deemed at risk of harm to themselves by the clinical team due to a sustained trajectory of recent weight loss.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Retention rate of participants at all five intervention sessions | 12 months
  At least 70% of those recruited will attend all 5 intervention sessions.
Number of eligible referrals that consent to participate | 12 months
  Over 50% of those who are referred to the study and are eligible to participate, will consent to take part in the study.
Proportion of missing data across outcome assessments | 12 months
  The level of missing data on clinical outcome measures at assessments (for those still retained in the study) does not exceed 20% per assessment
Adapted Experiences of Services Questionnaire | post-treatment (8 weeks).
  Adapted Experiences of Services Questionnaire measures satisfaction with experiences of therapy and will be used to gain feedback and measure aspects of the acceptability of the intervention. Seven items are rated on 0 to 3 scale, With higher item scores indicating greater satisfaction with therapy.

SECONDARY OUTCOMES:
The Eating Disorder Examination Questionnaire (EDE-Q) | post-treatment (8 weeks).
  A 28-item self-reported questionnaire adapted from the semi-structured interview Eating Disorder Examination (EDE) and designed to assess the range and severity of features associated with a diagnosis of eating disorder using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score. For each subscale scores range from 0 to 6, with higher scores indicating greater difficulties.
The Young Person's Clinical Outcome in Routine Evaluation (YP-CORE) | post-treatment (8 weeks). Follow-up (10 weeks)
  A 10-item questionnaire that measures psychological distress in young people. An evaluation of the YP-CORE showed good internal reliability and reliable change indices. Scorers range from 0 to 40, with higher scores indicating greater difficulties.
Recovery Questionnaire (ReQuest-YP) | post-treatment (8 weeks). Follow-up (10 weeks)
  Examines recovery of functionality and outlook post-treatment. An evaluation of the psychometric properties of the ReQuest-YP with 65 young people showed good internal consistency and test-retest reliability. Scores range from 0 to 90, with higher scores indicating greater recovery.
University of Rode Island Change Assessment Scale (URICA) | post-treatment (8 weeks). Follow-up (10 weeks)
  Examines a person's motivation to change in relation to a specific 'problem'. It is a 32-item self-report measure that includes 4 subscales to measure what stage of change the individual is currently in: Precontemplation, Contemplation, Action, and Maintenance. The scale consists of 4 subscales, each with scores ranging from 1 to 5, greater scores indicating greater motivation for change.
Repertory grid | post-treatment (8 weeks)
  Repertory grids are a type of interview tool which will be used to explore how participants perceive themselves and others in their lives. This will be developed with the participant prior to the intervention, to get a sense of their relational patterns at baseline. The grid will be developed using established techniques. Participants will then complete the same grid following the intervention to explore any changes in their perceptions of themselves and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Manchester Mental Health NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Given the small scale of the project there is no plan to make data available via online repositories. Anonymised data may be made available to other researchers on reasonable request.

REFERENCES:
- [Derived] Green C, Mannion G, Gill I, Hartley S, Dunlop BJ, Taylor PJ. Brief Cognitive Analytic Therapy (CAT)-Informed Reformulation for Young People With Eating Disorders: A Case Series. Clin Psychol Psychother. 2025 Mar-Apr;32(2):e70043. doi: 10.1002/cpp.70043. PMID 40171882